CLINICAL TRIAL: NCT05563324
Title: Genetics of Self-injurious Behaviour
Status: Completed | Type: Observational
Sponsor: University Medical Centre Maribor (Other)
Collaborators: Faculty of Medicine, University of Maribor (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRP-2013/01-07
Record Dates: First submitted 2022-05-03; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Self Injurious Behavior Without Suicidal Intent; Self-Injurious Behavior
Keywords: Self-Injurious Behavior; genetic polymorphisms; TPH1; SLC6A4; OPRM1; GNβ3; DRD2/ANKK1; anxiety; borderline personality disorder; trauma; impulsivity
MeSH Terms: conditions — Self-Injurious Behavior; Anxiety Disorders; Borderline Personality Disorder; Wounds and Injuries; Impulsive Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA isolated from whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- clinical sample: adolescents with nonsuicidal self-injury
  Interventions: Genetic: DNA extraction and genotyping of candidate genetic polymorphisms; Other: self-assessment questionnaires
- original control group: adolescents with no history of nonsuicidal self-injury
  Interventions: Genetic: DNA extraction and genotyping of candidate genetic polymorphisms; Other: self-assessment questionnaires
- general control group: adolescents from the general population
  Interventions: Genetic: DNA extraction and genotyping of candidate genetic polymorphisms

INTERVENTIONS:
Genetic: DNA extraction and genotyping of candidate genetic polymorphisms
Other: self-assessment questionnaires
  Groups: clinical sample; original control group

SUMMARY:
Nonsuicidal Self-Injury (NSSI) is being increasingly regarded as a separate psychiatric disorder. Since the latest Diagnostic and Statistical Manual of Mental Disorders - DSM-5 from 2013 defined NSSI as a separate diagnosis under section III - Conditions for Further Study, the knowledge about this field has increased considerably; however, the aetiology of this behaviour has still not been explained. There are many psychological explanations for the development and the continuation of NSSI. Researchers have identified the most common comorbidities (depression, borderline personality disorder, anxiety). The causes of NSSI are not known, although studies that have been carried out so far indicate both genetic and environmental factors.

The research included 95 adolescents with NSSI (participants were diagnosed based on the DSM-5 criteria), an original control group consisting of 21 people without NSSI, and 118 individuals from the general population as an additional control group for genetic research. For all participants we carried out the genotyping of polymorphisms for the TPH1 (rs4537731, rs1799913, rs7933505), SLC6A4 (VNTR STin2), OPRM1 (rs1799971), GNβ3 (rs5443) and DRD2/ANKK1 (rs1800497) genes. The participants with NSSI and the control group without NSSI completed translated questionnaires for the Barratt Impulsiveness Scale (BIS-11), State-Trait Anxiety Inventory for Adults (STAI), MacLean Screening Instrument for BPD (MSI-BPD) and the Early Trauma Inventory Self Report-Short Form (ETISR-SF). The participants with NSSI also completed the questionnaire for the Inventory of Statements about Self-Injury (ISAS), and the Self-Injury Craving Questionnaire (SICQ). The investigators carried out an association analysis and G x E analyses.

The aim of the research was to carry out the first G x E study on the etiology of NSSI in Slovene adolescents. We have hypothesized that NSSI could be associated with one of the candidate polymorphisms or a combination of candidate polymorphisms. Further we have hypothesized that the genetic polymorphisms associated to NSSI are the most connected to NSSI in traumatised individuals and that NSSI is associated with higher impulsivity.

DETAILED DESCRIPTION:
Theoretical background The etiology of Nonsuicidal Self-Injury (NSSI) has still not been explained. Studies that have been carried out so far indicate both genetic and environmental factors. It has been suggested, that NSSI is a polygenic disorder. Two neurotransmitter systems, the serotonergic system and the endogen opioids system, are the main candidate systems in the etiology of NSSI.

The serotonin system is important in comorbid disorders of NSSI (depression, anxiety…). There is also growing importance of its direct involvement in NSSI. Deficiency of tryptophan, a precursor of serotonin, has been connected with increasing frequency of NSSI. Variable-number tandem repeat polymorphism of the serotonin transporter gene - SLC6A4 (VNTR STin2) has been associated with borderline personality disorder, a disorder with frequent NSSI, in one study. The are some important polymorphisms of the gene for the tryptophan hydroxylase enzyme, the main enzyme in the synthesis of serotonin. The polymorphism rs1799913 has been associated with depression and with parasuicidal behavior. This polymorphism is, together with some other polymorphisms (e.g. rs4537731, rs7933505), a part of a haplotype. This haplotype has already shown some connections with borderline personality disorder.

There is also growing evidence that the changes in concentration of endogenous opioids (EO) could be associated with NSSI. Significantly lower β-endorphin and met-enkephalin values in the liquor of individuals with NSSI had been demonstrated. A recent study has shown significantly lower basal β-endorphin levels in adolescents with NSSI, when compared to healthy controls. Naomi I. Eisenberger is a leader in studying polymorphisms of endogenous opioids in conjunction with "emotional" pain. People with a lower threshold for physical pain also described a greater sensitivity to emotional pain. There is numerous evidence of the significant effect of the polymorphism of the gene for the mu-opioid receptor OPRM1 (A118G; rs1799971) on altered sensitivity to physical pain, pain perception and response to opiate analgesics. A significantly increased sensitivity of G allele carriers to social rejection (i.e. on a model for "emotional" pain) has been demonstrated. A number of studies have been conducted on the impact of the rs1799971 polymorphism on craving and addiction. Given the theoretical addictive background of NSSI and the interconnectedness of physical and emotional pain and the role of the rs1799971 polymorphism, this polymorphism is an important candidate polymorphism in NSSI. For individual addictions, different, partly conflicting results appear. Various studies have confirmed the G allele as a risk factor for various addictions, while others have not demonstrated any impact or have found a reduced risk of addiction in G allele carriers. Thus, in 2016, the first collaborative analysis was carried out in which 9064 subjects of the Caucasian population were included. In this large, European sample, the G allele proved to be a significant (OR = 0.90; confidence interval 95 % (0.83 - 0.97); p = 0.0095) protective factor for addiction in general. Direct studies of craving and the impact of rs1799971 on craving are rare and contradictory. There has been little research on potential genetic influences on the development of NSSI and rs1799971 does not appear to have been studied in this field.

The main target of antipsychotics, the dopamine receptor D2, is also important in the research of addiction. The most famous polymorphism of the dopamine receptor 2 gene is the Taq1A (TaqIA) (rs1800497) polymorphism. Two alleles of rs1800497 are known - A1 and A2. Allele A1 has been associated with pathological gambling, a typical behavioral addiction, in one study. It has also been associated with impulsivity and addictive behavior in some other studies. The A1 allele has also been associated with borderline personality traits. G - proteins have been connected with the proper activity of numerous receptors. The polymorphism C825T (rs5443) of the G protein beta 3 gene (GNbeta3) has in some research been connected with depression. In one study, the T allele carriers had a statistical higher risk for NSSI as other depressive patients.

Diminished pain perception and a higher pain threshold in people with NSSI have been shown.

Ethics committee approval and project registration The study has been approved by the Medical Ethics Committee of the Republic of Slovenia (number 69/06/13). It has been chosen and registered as an internal scientific research and developmental project of the University Medical Centre Maribor, Slovenia, on 1.8.2013 (project number IRP-2013/01-07).

Questionnaires All adolescents from the clinical sample and the original control group filled out the Slovenian version of the self-assessment questionnaire of the State-Trait Anxiety Inventory for Adults (STAI) and the following questionnaires, translated into Slovene: Barratt Impulsiveness Scale (BIS-11), MacLean Screening Instrument for BPD (MSI-BPD), Early Trauma Inventory Self Report-Short Form (ETISR-SF). The STAI measures two forms of anxiety. "State anxiety" measures the current state, i.e. the level of anxiety that the individual feels at a given event. "Trait anxiety" refers to the long-term state of the individual. BIS-11 is probably the most frequently used instrument for the measurement of impulsivity. The MSI-BPD is a screening questionnaire used to search for borderline personality disorder in adolescence. ETISR-SF measures the childhood trauma, including physical, emotional and sexual abuse, as well as general traumatic events.

In order to identify NSSI, the investigators used the Slovenian translation of the Inventory of Statements about Self-Injury (ISAS) and the Slovenian translation of the Self-Injury Craving Questionnaire (SICQ) for the clinical sample. The ISAS is a questionnaire consisting of two parts. The first part consists of 12 questions about self-injurious behavior and the second part of questions about 13 functions of NSSI. The SICQ contains 7 questions about the craving for NSSI.

DNA extraction and genotyping There is little research about genetics of NSSI. Some candidate genetic polymorphisms had been chosen with the help of this information. Predominantly, the candidate genetic polymorphisms in the study have therefor been chosen with the help of information about genetics of addiction and comorbid disorders (depression, borderline personality disorder, …).

DNA for genotyping was extracted from peripheral blood mononuclear cells using TRI-reagent (Sigma, Steinheim, Germany) according to manufacturer's instructions. Quality and concentration of extracted DNA was checked using agarose gel electrophoresis and SynergyTM 2 (Biotek, Winooski, VT, USA) spectrophotometer.

For the genotyping of the polymorphisms, the investigators first performed the real-time polymerase chain reaction (qPCR) and then the high resolution melting (HRM) or the restriction fragment length polymorphism (RFLP) method. The qPCR was performed as follows: denaturation at 95 °C for 10 min, multiplication, 45 cycles of 95°C 10 s, 60°C 15 s, 72°C 10 s. The HRM has been made at the following protocol: 95°C 1 min, 40°C 1 min, 60 - 90°C at 0,02 °C/s and cooling at 40°C for 10 s. The HRM reaction has been made with the LightCycler® 480 (Roche) and the LC480 HRM Master Mix (Roche) has been used. The investigators have analyzed the genotypes from the melting curves (TABLE 1). In the RFLP protocol, the product of the qPCR has been incubated with the right restriction enzyme from New England Biolabs (TABLE 1). Analysis has been done with agarose gel electrophoresis (2 % agarose gel, tris borate EDTA buffer). The DNA samples were mixed with 0.25% xylene cyanol and 40% sucrose. Electrophoresis has been run at 150 V for 20 minutes. At the end, the agarose gel has been analyzed under the UV light.

Gene; genetic polymorphism; sequence of the primer; temperature; genotyping method; restriction enzyme:

1. OPRM1; rs1799971; CGGTTCCTGGGTCAACTTGT, GATCGTGATGGCCGTGAT; 60 °C; HRM; /.
2. TPH1; rs4537731; GTTTCATGCAGGTATTAGTG, TGGCATTGAAGTAAGAGCAC; 60 °C; RFLP; Sau3AI.
3. TPH1; rs1799913; GTTAAGCACTGCAGCGTGAC, AAGCGGGACATGACCTAAGA; 60 °C; HRM; /.
4. TPH1; rs7933505; AAACTGAGAGGAAAATGCTTGC, CATTGCCGTTGAACTTTTGA; 65 °C; RFLP; NlaIII.
5. DRD2; rs1800497; CTTGCCCTCTAGGAAGGACAT, ACCTTCCTGAGTGTCATCAACC; 65 °C; RFLP; TaqI.
6. GNB3; rs5443; CATCATCTGCGGCATCACG, ACGCTCAGACTTCATGGAGT; 60 °C; HRM; /.
7. SLC6A4; VNTR; GGGCAATGTCTGGCGCTTCCCCTACATA, TTCTGGCCTCTCAAGAGGACCTACAGC; 65,5 °C; PCR; /.

Statistical analysis The data was analyzed using IBM SPSS Statistics program package (IMB Inc., Armonk, New York). P ≤ 0.05 was considered as statistically significant.

The comparison of the share of traumatized and abused adolescents in the clinical sample and in the original control group has been done with the Fisher's exact test. All continuous variables were first assessed for the normality using Kolmogorov-Smirnov test of normality. Correlation between the age at the onset of NSSI and the total number of NSSI in life was determined using Spearman's correlation. The relationship between the total number of self-injuries (NSSI) in life and the value on the SICQ questionnaire has also been assessed using Spearman's correlation analysis. Relationship of the value of the SICQ questionnaire and the time that passes from the thought of NSSI to NSSI and also genotype and the total number of NSSI in life both have been assessed using Kruskal-Wallis H-test. The Mann-Whitney U-test had been used to determine the relationship between genotype and the age at the onset of NSSI. Different logistic regression models with parameters of the ETISR-SF questionnaire / BIS-11 / MSI - BPD / STAI STETE / STAI TRAIT and the candidate genotypes as independent variables and NSSI as dependent variable have been made. Unadjusted analyses of the rs1799971 / rs1800497 genotype itself and craving variable were carried out using Mann-Whitney U-test. The contribution of the rs1799971 / rs1800497 genotype to the level of craving for NSSI (SICQ) was studied using generalized linear models and was adjusted to STAI STATE and STAI TRAIT / ETISR - SF. Logistic regression models with candidate genotypes as independent variables and pain perception during NSSI as dependent variable have been made. The contribution of the rs1799971 / rs1800497 genotype to pain perception has been studied using logistic regression models that were adjusted to STAI STATE / STAI TRAIT / MSI - BPD/ ETISR - SF. The relationship between pain perception during NSSI and craving (SICQ) was assessed using Mann-Whitney U-test.

Aim of the study and the hypotheses The aim of the research was to carry out the first G x E study on the etiology of NSSI, diagnosed with the proposed research criteria from DSM-5, in Slovene adolescents. The investigators wanted to make the first association study of the rs1799971 in adolescents with NSSI and study the connection of the OPRM1 gene with addictive properties of NSSI and craving for NSSI. The goal was also to replicate the results of Joyce and his colleges (association of rs5443 and NSSI in depressive patients) in a sample of adolescents with NSSI.

The investigators have hypothesized that NSSI could be associated with one of the candidate polymorphisms or a combination of candidate polymorphisms. Further the investigators have hypothesized that the genetic polymorphisms associated to NSSI are the most connected to NSSI in traumatised individuals and that NSSI is associated with higher impulsivity.

ELIGIBILITY:
Clinical sample

Inclusion Criteria

All of the adolescents from the clinical sample met the research criteria for NSSI proposed in section III (Conditions for further study) of the DSM-5 (American Psychiatric Association, 2013):

(A)In the last year, the individual has, on 5 or more days, engaged in intentional self-inflicted damage to the surface of his or her body of a sort likely to induce bleeding, bruising, or pain (e.g., cutting, burning, stabbing, hitting, and excessive rubbing), with the expectation that the injury will lead to only minor or moderate physical harm (i.e., there is no suicidal intent). Note: The absence of suicidal intent has either been stated by the individual or can be inferred by the individual's repeated engagement in a behavior that the individual knows, or has learned, is not likely to result in death.

(B)The individual engages in the self-injurious behavior with one or more of the following expectations:(1)to obtain relief from a negative feeling or cognitive state,(2)to resolve an interpersonal difficulty,(3)to induce a positive feeling state. Note: The desired relief or response is experienced during or shortly after the self-injury, and the individual may display patterns of behavior suggesting a dependence on repeatedly engaging in it.

(C)The intentional self-injury is associated with at least one of the following:(1)interpersonal difficulties or negative feelings or thoughts, such as depression, anxiety, tension, anger, generalized distress, or self-criticism, occurring in the period immediately prior to the self-injurious act,(2)prior to engaging in the act, a period of preoccupation with the intended behavior that is difficult to control,(3)thinking about self-injury that occurs frequently, even when it is not acted upon.

(D)The behavior is not socially sanctioned (e.g., body piercing, tattooing, part of a religious or cultural ritual) and is not restricted to picking a scab or nail biting.

(E)The behavior or its consequences cause clinically significant distress or interference in interpersonal, academic, or other important areas of functioning.

(F)The behavior does not occur exclusively during psychotic episodes, delirium, substance intoxication, or substance withdrawal. In individuals with a neurodevelopmental disorder, the behavior is not part of a pattern of repetitive stereotypies. The behavior is not better explained by another mental disorder or medical condition (e.g., psychotic disorder, autism spectrum disorder, intellectual disability, Lesch-Nyhan syndrome, stereotyped movement disorder with self-injury, trichotillomania [hair pulling disorder], and excoriation [skin picking disorder]).

Exclusion Criteria Criterion F of the research criteria for NSSI is a exclusion criterion and has been used as such also in our research.

Control group

Inclusion Criteria:

* absence of NSSI behavior over a lifetime,
* no treatment by a psychologist or a (child and adolescent) psychiatrist ever in life,
* age between 12 and 21 years.

Exclusion Criteria:

* a diagnosis of mental disorder,
* intellectual disability,
* autism spectrum disorder.

General control group

Inclusion Criteria:

- age between 18 and 24 years.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Clinical sample We have invited 96 adolescents (12 - 21 years) with NSSI to participate in our study. The adolescents have been patients of the Paediatrics Clinic - University Clinical Centre Maribor, or the Unit for Adolescent Psychiatry - University Psychiatric Clinic Ljubljana, or the Child and adolescent Psychiatry - Health Care Centre Dr Adolf Drolc Maribor or have been treated by Natasa Potocnik Dajcman, M.D.. DNA of 95 adolescents could be isolated properly.
  Control group We have invited 96 adolescents (12 - 21 years) with no history of NSSI. From those adolescents, we managed to create an original control group with 21 participants.
  General control group Because of the demands of the genetics analysis, we have formed one more control group - the general control group. This control group was formed from 118 adolescents (18- 24 years) of the general population, that donated their DNA samples for research purposes.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2014-05-09 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-06-18 (Actual)

PRIMARY OUTCOMES:
Two generalized linear models between the polymorphism rs1799971 of the OPRM1 gene, two types of anxiety as covariates and craving for NSSI as dependent variable. | All of the included parameters are a one time measure.
  The two types of anxiety measured with State-Trait Anxiety Inventory for Adults (STAI), which measures "State anxiety" - i.e. the level of anxiety that the individual feels at a given event and "Trait anxiety" - long-term state of the individual. Craving measured with Self-Injury Craving Questionnaire (SICQ).
A logistic regression with the overall Early Trauma Inventory Self Report-Short Form (ETISR-SF) score, as well as SLC6A4 VNTR status as independent variables and the presence of NSSI as a dependent variable. | All of the included parameters are a one time measure.
  The presence of NSSI has been determined with the group status (clinical sample or control group) of the participant.
Measurement of the craving for NSSI (with the Self-Injury Craving Questionnaire score) for the participants in the clinical sample. | All of the included parameters are a one time measure.
  Calculation of the average craving for NSSI in the clinical sample has been made. Comparison of the average craving for NSSI in the clinical sample with the average cocaine craving score from the reference article has been made.
A logistic regression with the overall Early Trauma Inventory Self Report-Short Form (ETISR-SF) score, as well as rs1800497 polymorphism status as independent variables and the presence of NSSI as a dependent variable. | All of the included parameters are a one time measure.
  The presence of NSSI has been determined with the group status (clinical sample or control group) of the participant.
Analysis of the relationship between candidate genotypes and pain perception during NSSI. | All of the included parameters are a one time measure.
  Logistic regression models with candidate genotypes as independent variables and pain perception during NSSI as dependent variable have been made. The contribution of the rs1799971 / rs1800497 genotype to pain perception has been studied using logistic regression models that were adjusted to STAI STATE / STAI TRAIT / MSI - BPD/ ETISR - SF.

SECONDARY OUTCOMES:
Analysis of the relationship between rs4537731 polymorphism status of the TPH 1 gene and age at the beginning of NSSI. | All of the included parameters are a one time measure.
  Age at the beginning of NSSI has been measured with the Inventory of Statements about Self - Injury. In statistical analysis the Mann - Whitney U-test has been used.
Analysis of the relationship between craving for NSSI as measured by Self-Injury Craving Questionnaire score and the number of NSSI episodes during lifetime (measured with the Inventory of Statements about Self - Injury). | All of the included parameters are a one time measure.
Different logistic regression models with parameters of the ETISR-SF / BIS-11 / MSI - BPD / STAI STETE / STAI TRAIT and rs5443 (GNβ3 gene) as independent variable and NSSI as dependent variable have been made. | All of the included parameters are a one time measure.

OTHER OUTCOMES:
Analysis of the relationship between trauma and abuse, measured by the Early Trauma Inventory Self Report-Short Form (ETISR-SF), and NSSI. | All of the included parameters are a one time measure.
  Fisher´s exact test between ETISR-SF (traumatized or not according to overall score, emotional / sexual / physical abused or nor, general trauma in childhood or not) in the clinical sample and in the original control group.

CONTACTS AND LOCATIONS:
Overall Officials: Hojka Gregorič Kumperščak, M.D., Ph.D., Study Director — University Medical Centre Maribor and Faculty of Medicine, University of Maribor; Uroš Potočnik, Ph.D., Study Chair — Faculty of Medicine, University of Maribor; Teja Bunderla, M.D., Ph.D., Principal Investigator — at the time of research - University Medical Centre Maribor, now - Gesellschaft zur Förderung seelischer Gesundheit GmbH

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan to share the IPD systematically yet, but there are also no reasons, why it would not be shared. If there is interest, IPD could be shared.

REFERENCES:
- [Background] McCloskey MS, Ben-Zeev D, Lee R, Berman ME, Coccaro EF. Acute tryptophan depletion and self-injurious behavior in aggressive patients and healthy volunteers. Psychopharmacology (Berl). 2009 Mar;203(1):53-61. doi: 10.1007/s00213-008-1374-6. Epub 2008 Oct 23. PMID 18946662
- [Background] Ni X, Chan K, Bulgin N, Sicard T, Bismil R, McMain S, Kennedy JL. Association between serotonin transporter gene and borderline personality disorder. J Psychiatr Res. 2006 Aug;40(5):448-53. doi: 10.1016/j.jpsychires.2006.03.010. Epub 2006 May 11. PMID 16690085
- [Background] Jokela M, Raikkonen K, Lehtimaki T, Rontu R, Keltikangas-Jarvinen L. Tryptophan hydroxylase 1 gene (TPH1) moderates the influence of social support on depressive symptoms in adults. J Affect Disord. 2007 Jun;100(1-3):191-7. doi: 10.1016/j.jad.2006.10.016. Epub 2006 Nov 28. PMID 17134762
- [Background] Gizatullin R, Zaboli G, Jonsson EG, Asberg M, Leopardi R. Haplotype analysis reveals tryptophan hydroxylase (TPH) 1 gene variants associated with major depression. Biol Psychiatry. 2006 Feb 15;59(4):295-300. doi: 10.1016/j.biopsych.2005.07.034. Epub 2005 Sep 13. PMID 16165107
- [Background] Zaboli G, Gizatullin R, Nilsonne A, Wilczek A, Jonsson EG, Ahnemark E, Asberg M, Leopardi R. Tryptophan hydroxylase-1 gene variants associate with a group of suicidal borderline women. Neuropsychopharmacology. 2006 Sep;31(9):1982-90. doi: 10.1038/sj.npp.1301046. Epub 2006 Feb 22. PMID 16495936
- [Background] Stanley B, Sher L, Wilson S, Ekman R, Huang YY, Mann JJ. Non-suicidal self-injurious behavior, endogenous opioids and monoamine neurotransmitters. J Affect Disord. 2010 Jul;124(1-2):134-40. doi: 10.1016/j.jad.2009.10.028. Epub 2009 Nov 25. PMID 19942295
- [Background] van der Venne P, Balint A, Drews E, Parzer P, Resch F, Koenig J, Kaess M. Pain sensitivity and plasma beta-endorphin in adolescent non-suicidal self-injury. J Affect Disord. 2021 Jan 1;278:199-208. doi: 10.1016/j.jad.2020.09.036. Epub 2020 Sep 11. PMID 32961416
- [Background] Eisenberger NI, Jarcho JM, Lieberman MD, Naliboff BD. An experimental study of shared sensitivity to physical pain and social rejection. Pain. 2006 Dec 15;126(1-3):132-8. doi: 10.1016/j.pain.2006.06.024. Epub 2006 Aug 4. PMID 16890354
- [Background] Eisenberger NI. Why rejection Hurts: What Social Neuroscience Has Revealed abaut the Brain's Response to Social rejection. Future Science: Essays from the Cutting Edge. 2011; 39: 586-598.
- [Background] Eisenberger NI. The neural bases of social pain: evidence for shared representations with physical pain. Psychosom Med. 2012 Feb-Mar;74(2):126-35. doi: 10.1097/PSY.0b013e3182464dd1. Epub 2012 Jan 27. PMID 22286852
- [Background] Klepstad P, Rakvag TT, Kaasa S, Holthe M, Dale O, Borchgrevink PC, Baar C, Vikan T, Krokan HE, Skorpen F. The 118 A > G polymorphism in the human mu-opioid receptor gene may increase morphine requirements in patients with pain caused by malignant disease. Acta Anaesthesiol Scand. 2004 Nov;48(10):1232-9. doi: 10.1111/j.1399-6576.2004.00517.x. PMID 15504181
- [Background] Chou WY, Yang LC, Lu HF, Ko JY, Wang CH, Lin SH, Lee TH, Concejero A, Hsu CJ. Association of mu-opioid receptor gene polymorphism (A118G) with variations in morphine consumption for analgesia after total knee arthroplasty. Acta Anaesthesiol Scand. 2006 Aug;50(7):787-92. doi: 10.1111/j.1399-6576.2006.01058.x. PMID 16879459
- [Background] Walter C, Doehring A, Oertel BG, Lotsch J. micro-opioid receptor gene variant OPRM1 118 A>G: a summary of its molecular and clinical consequences for pain. Pharmacogenomics. 2013 Nov;14(15):1915-25. doi: 10.2217/pgs.13.187. PMID 24236490
- [Background] Matic M, de Wildt SN, Tibboel D, van Schaik RHN. Analgesia and Opioids: A Pharmacogenetics Shortlist for Implementation in Clinical Practice. Clin Chem. 2017 Jul;63(7):1204-1213. doi: 10.1373/clinchem.2016.264986. PMID 28637770
- [Background] Way BM, Taylor SE, Eisenberger NI. Variation in the mu-opioid receptor gene (OPRM1) is associated with dispositional and neural sensitivity to social rejection. Proc Natl Acad Sci U S A. 2009 Sep 1;106(35):15079-84. doi: 10.1073/pnas.0812612106. Epub 2009 Aug 14. PMID 19706472
- [Background] Schinka JA, Town T, Abdullah L, Crawford FC, Ordorica PI, Francis E, Hughes P, Graves AB, Mortimer JA, Mullan M. A functional polymorphism within the mu-opioid receptor gene and risk for abuse of alcohol and other substances. Mol Psychiatry. 2002;7(2):224-8. doi: 10.1038/sj.mp.4000951. PMID 11840318
- [Background] Coller JK, Beardsley J, Bignold J, Li Y, Merg F, Sullivan T, Cox TC, Somogyi AA. Lack of association between the A118G polymorphism of the mu opioid receptor gene (OPRM1) and opioid dependence: A meta-analysis. Pharmgenomics Pers Med. 2009;2:9-19. Epub 2009 Mar 20. PMID 23226031
- [Background] Chen D, Liu L, Xiao Y, Peng Y, Yang C, Wang Z. Ethnic-specific meta-analyses of association between the OPRM1 A118G polymorphism and alcohol dependence among Asians and Caucasians. Drug Alcohol Depend. 2012 Jun 1;123(1-3):1-6. doi: 10.1016/j.drugalcdep.2011.10.012. Epub 2011 Nov 8. PMID 22071118
- [Background] Koller G, Zill P, Rujescu D, Ridinger M, Pogarell O, Fehr C, Wodarz N, Bondy B, Soyka M, Preuss UW. Possible association between OPRM1 genetic variance at the 118 locus and alcohol dependence in a large treatment sample: relationship to alcohol dependence symptoms. Alcohol Clin Exp Res. 2012 Jul;36(7):1230-6. doi: 10.1111/j.1530-0277.2011.01714.x. Epub 2012 Feb 6. PMID 22309038
- [Background] Haerian BS, Haerian MS. OPRM1 rs1799971 polymorphism and opioid dependence: evidence from a meta-analysis. Pharmacogenomics. 2013 May;14(7):813-24. doi: 10.2217/pgs.13.57. PMID 23651028
- [Background] Woodcock EA, Lundahl LH, Burmeister M, Greenwald MK. Functional mu opioid receptor polymorphism (OPRM1 A(118) G) associated with heroin use outcomes in Caucasian males: A pilot study. Am J Addict. 2015 Jun;24(4):329-35. doi: 10.1111/ajad.12187. Epub 2015 Apr 24. PMID 25911999
- [Background] Lechner WV, Knopik VS, McGeary JE, Spillane NS, Tidey JW, McKee SA, Metrik J, Leventhal AM, Rohsenow DJ, Kahler CW. Influence of the A118G Polymorphism of the OPRM1 Gene and Exon 3 VNTR Polymorphism of the DRD4 Gene on Cigarette Craving After Alcohol Administration. Nicotine Tob Res. 2016 May;18(5):632-6. doi: 10.1093/ntr/ntv136. Epub 2015 Jun 19. PMID 26092968
- [Background] Sloan ME, Klepp TD, Gowin JL, Swan JE, Sun H, Stangl BL, Ramchandani VA. The OPRM1 A118G polymorphism: converging evidence against associations with alcohol sensitivity and consumption. Neuropsychopharmacology. 2018 Jun;43(7):1530-1538. doi: 10.1038/s41386-017-0002-8. Epub 2018 Feb 2. PMID 29497164
- [Background] Bach P, Weil G, Pompili E, Hoffmann S, Hermann D, Vollstadt-Klein S, Mann K, Perez-Ramirez U, Moratal D, Canals S, Dursun SM, Greenshaw AJ, Kirsch P, Kiefer F, Sommer WH. Incubation of neural alcohol cue reactivity after withdrawal and its blockade by naltrexone. Addict Biol. 2020 Jan;25(1):e12717. doi: 10.1111/adb.12717. Epub 2019 Feb 12. PMID 30748046
- [Background] Schwantes-An TH, Zhang J, Chen LS, Hartz SM, Culverhouse RC, Chen X, Coon H, Frank J, Kamens HM, Konte B, Kovanen L, Latvala A, Legrand LN, Maher BS, Melroy WE, Nelson EC, Reid MW, Robinson JD, Shen PH, Yang BZ, Andrews JA, Aveyard P, Beltcheva O, Brown SA, Cannon DS, Cichon S, Corley RP, Dahmen N, Degenhardt L, Foroud T, Gaebel W, Giegling I, Glatt SJ, Grucza RA, Hardin J, Hartmann AM, Heath AC, Herms S, Hodgkinson CA, Hoffmann P, Hops H, Huizinga D, Ising M, Johnson EO, Johnstone E, Kaneva RP, Kendler KS, Kiefer F, Kranzler HR, Krauter KS, Levran O, Lucae S, Lynskey MT, Maier W, Mann K, Martin NG, Mattheisen M, Montgomery GW, Muller-Myhsok B, Murphy MF, Neale MC, Nikolov MA, Nishita D, Nothen MM, Nurnberger J, Partonen T, Pergadia ML, Reynolds M, Ridinger M, Rose RJ, Rouvinen-Lagerstrom N, Scherbaum N, Schmal C, Soyka M, Stallings MC, Steffens M, Treutlein J, Tsuang M, Wall TL, Wodarz N, Yuferov V, Zill P, Bergen AW, Chen J, Cinciripini PM, Edenberg HJ, Ehringer MA, Ferrell RE, Gelernter J, Goldman D, Hewitt JK, Hopfer CJ, Iacono WG, Kaprio J, Kreek MJ, Kremensky IM, Madden PA, McGue M, Munafo MR, Philibert RA, Rietschel M, Roy A, Rujescu D, Saarikoski ST, Swan GE, Todorov AA, Vanyukov MM, Weiss RB, Bierut LJ, Saccone NL. Association of the OPRM1 Variant rs1799971 (A118G) with Non-Specific Liability to Substance Dependence in a Collaborative de novo Meta-Analysis of European-Ancestry Cohorts. Behav Genet. 2016 Mar;46(2):151-69. doi: 10.1007/s10519-015-9737-3. Epub 2015 Sep 21. PMID 26392368
- [Background] Kaess M, Hooley JM, Klimes-Dougan B, Koenig J, Plener PL, Reichl C, Robinson K, Schmahl C, Sicorello M, Westlund Schreiner M, Cullen KR. Advancing a temporal framework for understanding the biology of nonsuicidal self- injury: An expert review. Neurosci Biobehav Rev. 2021 Nov;130:228-239. doi: 10.1016/j.neubiorev.2021.08.022. Epub 2021 Aug 24. PMID 34450182
- [Background] Neville MJ, Johnstone EC, Walton RT. Identification and characterization of ANKK1: a novel kinase gene closely linked to DRD2 on chromosome band 11q23.1. Hum Mutat. 2004 Jun;23(6):540-5. doi: 10.1002/humu.20039. PMID 15146457
- [Background] Grandy DK, Litt M, Allen L, Bunzow JR, Marchionni M, Makam H, Reed L, Magenis RE, Civelli O. The human dopamine D2 receptor gene is located on chromosome 11 at q22-q23 and identifies a TaqI RFLP. Am J Hum Genet. 1989 Nov;45(5):778-85. PMID 2573278
- [Background] Eisenberg DT, Mackillop J, Modi M, Beauchemin J, Dang D, Lisman SA, Lum JK, Wilson DS. Examining impulsivity as an endophenotype using a behavioral approach: a DRD2 TaqI A and DRD4 48-bp VNTR association study. Behav Brain Funct. 2007 Jan 10;3:2. doi: 10.1186/1744-9081-3-2. PMID 17214892
- [Background] White MJ, Morris CP, Lawford BR, Young RM. Behavioral phenotypes of impulsivity related to the ANKK1 gene are independent of an acute stressor. Behav Brain Funct. 2008 Nov 24;4:54. doi: 10.1186/1744-9081-4-54. PMID 19025655
- [Background] Comings DE, Rosenthal RJ, Lesieur HR, Rugle LJ, Muhleman D, Chiu C, Dietz G, Gade R. A study of the dopamine D2 receptor gene in pathological gambling. Pharmacogenetics. 1996 Jun;6(3):223-34. doi: 10.1097/00008571-199606000-00004. PMID 8807661
- [Background] Noble EP. D2 dopamine receptor gene in psychiatric and neurologic disorders and its phenotypes. Am J Med Genet B Neuropsychiatr Genet. 2003 Jan 1;116B(1):103-25. doi: 10.1002/ajmg.b.10005. PMID 12497624
- [Background] Nemoda Z, Lyons-Ruth K, Szekely A, Bertha E, Faludi G, Sasvari-Szekely M. Association between dopaminergic polymorphisms and borderline personality traits among at-risk young adults and psychiatric inpatients. Behav Brain Funct. 2010 Jan 12;6:4. doi: 10.1186/1744-9081-6-4. PMID 20205808
- [Background] Lee HJ, Cha JH, Ham BJ, Han CS, Kim YK, Lee SH, Ryu SH, Kang RH, Choi MJ, Lee MS. Association between a G-protein beta 3 subunit gene polymorphism and the symptomatology and treatment responses of major depressive disorders. Pharmacogenomics J. 2004;4(1):29-33. doi: 10.1038/sj.tpj.6500217. PMID 14647404
- [Background] Cao MQ, Hu SY, Zhang CH, Xia DS. Study on the interrelationship between 5-HTTLPR/G-protein beta3 subunit (C825T) polymorphisms and depressive disorder. Psychiatr Genet. 2007 Aug;17(4):233-8. doi: 10.1097/YPG.0b013e3280c1e5de. PMID 17621167
- [Background] Lopez-Leon S, Janssens AC, Gonzalez-Zuloeta Ladd AM, Del-Favero J, Claes SJ, Oostra BA, van Duijn CM. Meta-analyses of genetic studies on major depressive disorder. Mol Psychiatry. 2008 Aug;13(8):772-85. doi: 10.1038/sj.mp.4002088. Epub 2007 Oct 16. PMID 17938638
- [Background] Joyce PR, McKenzie JM, Mulder RT, Luty SE, Sullivan PF, Miller AL, Kennedy MA. Genetic, developmental and personality correlates of self-mutilation in depressed patients. Aust N Z J Psychiatry. 2006 Mar;40(3):225-9. doi: 10.1080/j.1440-1614.2006.01778.x. PMID 16476149
- [Background] Noblin JL, Venta A, Sharp C. The validity of the MSI-BPD among inpatient adolescents. Assessment. 2014 Apr;21(2):210-7. doi: 10.1177/1073191112473177. Epub 2013 Jan 23. PMID 23344914
- [Background] Chanen AM, Jovev M, Djaja D, McDougall E, Yuen HP, Rawlings D, Jackson HJ. Screening for borderline personality disorder in outpatient youth. J Pers Disord. 2008 Aug;22(4):353-64. doi: 10.1521/pedi.2008.22.4.353. PMID 18684049
- [Background] Victor SE, Glenn CR, Klonsky ED. Is non-suicidal self-injury an "addiction"? A comparison of craving in substance use and non-suicidal self-injury. Psychiatry Res. 2012 May 15;197(1-2):73-7. doi: 10.1016/j.psychres.2011.12.011. Epub 2012 Mar 6. PMID 22401975
- [Background] Bunderla T, Kumperscak HG. Altered pain perception in self-injurious behavior and the association of psychological elements with pain perception measures: a systematic review. Psychiatr Danub. 2015 Dec;27(4):346-54. PMID 26609646
- [Background] Koenig J, Thayer JF, Kaess M. A meta-analysis on pain sensitivity in self-injury. Psychol Med. 2016 Jun;46(8):1597-612. doi: 10.1017/S0033291716000301. Epub 2016 Mar 11. PMID 26964517